CLINICAL TRIAL: NCT02165124
Title: Bariatric Embolization of Arteries for the Treatment of Obesity
Acronym: BEAT Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00093563
Record Dates: First submitted 2014-06-11; First posted 2014-06-17 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Morbid Obesity
Keywords: Obesity; Morbid Obesity; Bariatric Surgery; Embolization; Minimally Invasive; Weight Loss
MeSH Terms: conditions — Obesity, Morbid; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention/Bariatric Embolization (Experimental)
  Interventions: Device: Artificial Embolization Device

INTERVENTIONS:
Device: Artificial Embolization Device — Embosphere Microspheres
  Other Names: Device Product Codes: 85 NAJ; Classification Name: Artificial Embolization Device; Regulation Numbers: 21 CFR 882.5950

SUMMARY:
The purpose of this study is evaluate the safety and effectiveness of bariatric embolization as a minimally-invasive image-guided procedure for morbid obesity. In this procedure, specific blood vessels to the stomach are blocked in order to suppress some of the body's signals for feeling hungry, leading to weight loss.

Morbid obesity is currently treated with diet and exercise, medications, and surgery. This study is designed to help treat obesity using a minimally invasive, non-surgical, angiographic (through the blood vessel) approach. This procedure is similar to a common procedure used to treat bleeding within the stomach. This version of the procedure has been named "bariatric embolization".

Although there are over 40 hormones that limit food intake, there is only one hormone, ghrelin that has been shown to stimulate (prompt) food intake. In obese patients, eating fails to suppress ghrelin levels, which is believed to prevent feeling full after a meal and to lead to overeating. Due to the strong hunger craving effects of ghrelin, this hormone has been a target for the treatment of obesity and weight loss. More recently, ghrelin has been shown to have a significant role in the long-term effect of weight loss in bariatric (obesity) surgery where ghrelin levels are shown to be much lower when compared to untreated patients.

Recent data collected in animals in has shown that blocking blood vessels to a particular portion of the stomach (bariatric embolization) can temporarily decrease levels of the appetite inducing hormone ghrelin, and decrease short-term weight gain. In a study of 5 people, there was a decrease in ghrelin levels and weight loss in the first month after the procedure, but there is no information about the effects of the procedure over longer periods of time.

The investigator hopes to learn if bariatric embolization results in safe and effective weight loss in people who are morbidly obese.

ELIGIBILITY:
Inclusion Criteria:

1. Willing, able and mentally competent to provide written informed consent.
2. Body mass index (BMI) between 40-60.
3. Residence within 25 miles of the enrolling institution
4. Vascular anatomy (including celiac, hepatic, and gastric arteries) that in the opinion of the interventional radiologist amenable to Bariatric Embolization, as assessed on 3D CT angiography.
5. Suitable for protocol therapy as determined by the interventional radiology Investigator.
6. Adequate hematological, hepatic and renal function as follows:

   Hematological Neutrophils > 1.5 x 109/L Platelets > 100 x 109/L International Normalized Ratio (INR) <1.5

   Hepatic Bilirubin ≤ 2.0 mg/dL Albumin ≥ 2.5 g/L

   Renal Estimated Glomerular Filtration Rate (GFR) > 60ml/min.1.73m2
7. Aged 18 years or older.

Exclusion Criteria:

1. Prior history of gastric pancreatic, hepatic, and/or splenic surgery
2. Prior radiation to the upper abdomen
3. Prior embolization to the stomach, spleen or liver
4. Portal venous hypertension
5. Prior or current history of peptic ulcer disease
6. Hiatal Hernia
7. Significant risk factors for peptic ulcer disease including daily NSAID use and smoking.
8. Active H. Pylori infection
9. Weight greater than 400 pound
10. Known aortic pathology such as aneurysm or dissection renal insufficiency as evidenced by an estimated glomerular filtration rate of < 60 milliliters per minute
11. Major comorbidity such as cancer, significant cardiovascular disease, diabetes, or peripheral arterial disease.
12. Complicated arterial anatomic variants including left gastric artery arising from the aorta, and/or hepatic arterial supply via a replaced or accessory left hepatic artery arising from the left gastric artery.
13. Pregnancy
14. Preexisting chronic abdominal pain
15. Positive stool occult study
16. Abnormal Endoscopy
17. Abnormal Nuclear Gastric Motility examination
18. American Society of Anaesthesiologists (ASA) Class 4 or 5 (very high risk surgical candidates: class 4= incapacitating disease that is a constant threat to life) at the time of screening for enrollment into the study will be excluded from participation. This exclusion criterion exists because of the possibility that surgical intervention will be needed if the study intervention subsequently leads to severe adverse effects.
19. History of Inflammatory Bowel Disease
20. Autoimmune disease
21. Cirrhosis
22. Known history of allergy to iodinated contrast media

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifford R Weiss, M.D., Principal Investigator — Johns Hopkins University; Aravind Arepally, M.D., Principal Investigator — Piedmont Healthcare; Dara L Kraitchman, V.M.D., Ph.D., Principal Investigator — Johns Hopkins University; Lawrence Cheskin, M.D., Study Chair — Johns Hopkins University; Aaron Fischman, M.D, Principal Investigator — Icahn School of Medicine at Mount Sinai - aaron.fischman@mountsinai.org ; 212-241-7409; Ellen Weiss, B.S, M.A, M.S, Study Chair — Icahn School of Medicine at Mount Sinai - ellen.weiss@mountsinai.org ; 212-241-2317
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention/Bariatric Embolization
Started | 20
Completed | 15
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Intervention/Bariatric Embolization
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Percent Weight Change
Description: This will be assessed by Percentage of excess weight loss (EWL). Percentage of excess weight loss is calculated by measuring the participants excess weight at baseline and then calculating the percentage of excess weight that was lost 12 months after surgery (for example if a participant has 100 pounds of excess weight prior to surgery and loses 30 pounds, their excess weight loss would be 30%).
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: percentage of excess weight loss
Arm/Group | Intervention/Bariatric Embolization
Number analyzed (Participants) | 20
percentage of excess weight loss | 11.5 (10.2)

2. Other Pre Specified Outcome: Blood Pressure
Description: Unit of Measure: mmHg
Time Frame: 12 Months
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Lipid Panel
Description: Unit of Measure: mg/dL, Total cholesterol, High-density lipoprotein cholesterol (HDL-C) - often called "good cholesterol" , Low-density lipoprotein cholesterol (LDL-C) - often called "bad cholesterol" and Triglycerides
Time Frame: 12 Months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Ghrelin Levels
Description: Unit of Measure: pg/mL, Ghrelin on the other hand is a fast-acting hormone, seemingly playing a role in meal initiation.
Time Frame: 12 Months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Serum Obesity Hormone(Leptin)
Description: This will be assessed by Leptin concentration
  Unit of Measure: pg/mL, Leptin is a mediator of long-term regulation of energy balance, suppressing food intake and thereby inducing weight loss.
Time Frame: 12 Months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Eating and Hunger/Satiety Assessments
Description: Unit of Measure: N/A Utilizing 3-Factor Eating Questionnaire Scores
Time Frame: 12 Months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Quality of Life Parameters Survey
Description: Unit of Measure: N/A Utilizing Short Form Health Survey (SF)-36 and Impact of Weight on Quality of Life (IWQOL)-Lite
Time Frame: 12 Months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Food Intake
Description: Documented via journal entries
Time Frame: 12 Months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Results From Endoscopy
Description: Photos and clinical reports analyzed
Time Frame: 12 Months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Gastric Motility/Emptying
Description: Unit of Measure: (t 1/2) in minutes, A gastric emptying scan (GES) is a nuclear medicine exam that uses a radioactive material that you will eat in a meal. You will eat this meal in the Radiology department before your scan. The radioactive material allows doctors to see how your stomach empties.
  This scan is used to help diagnose conditions called motility disorders. These are conditions that change the way the stomach contracts and moves food into your intestines. A GES is a form of radiology, because radiation is used to take pictures of your body.
Time Frame: 12 Months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | Intervention/Bariatric Embolization
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 8/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention/Bariatric Embolization (N=20)
asymptomatic gastric ulcers discovered on endoscopy (Gastrointestinal disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT02165124/Prot_SAP_000.pdf